CLINICAL TRIAL: NCT02560129
Title: Evaluation of Outcomes Following Critical Illness Through a MICU Recovery Clinic
Brief Title: MICU Recovery Clinic
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00031295
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Sepsis; Respiratory Failure; ARDS
Keywords: recovery; ICU; clinic; survivor; physical function
MeSH Terms: conditions — Critical Illness; Sepsis; Respiratory Insufficiency | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU Survivors: ICU survivors will be seen in a MICU Recovery Clinic where Questionnaires, Physical and Cognitive Function assessments will be measured
  Interventions: Other: Questionnaires, Physical and Cognitive Function

INTERVENTIONS:
Other: Questionnaires, Physical and Cognitive Function — ICU survivors will be administered a battery of questionnaires. Measurements of physical and cognitive function will also be performed.

SUMMARY:
Summary: Emerging data demonstrate long-term morbidity and mortality in those who survive critical illness. However, there is no data regarding long-term follow-up for ICU survivors. The investigators have begun the implementation of an ICU recovery clinic.

Rationale:

ICU survivors are at high risk for functional, cognitive and psychiatric impairments. However, methods to mitigate these impairments and improve recovery are lacking. Special follow-up clinics for survivors of critical illness have been proposed and implemented to some degree, but are uncommon.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate physical function, cognitive function, and overall functional status during recovery from critical illness.
2. To evaluate anxiety, depression, and PTSD during recovery from critical illness.
3. To evaluate resilience during recovery from critical illness.
4. To evaluate healthcare utilization rates, morbidity, and mortality following critical illness.
5. Added April 2016: To study the voice and swallowing function of patients following recovery from critical illness.
6. Added April 2016: To study the pain of patients following recovery from critical illness.

Intervention:

A prospective observational study of all patients who attend our ICU recovery clinic.

Methods:

Patients will be identified for participation in our ICU Recovery Clinic during their admission to the Wake Forest Baptist Medical Center Medical Intensive Care Unit (MICU). They will be asked to return to the ICU recovery clinic within 1 month of hospital discharge. Structured clinic visits as standard of care will include medication reconciliation and evaluation by a pharmacist, along with an evaluation by a clinic physician to address acute medical issues and provide counselling. They will also undergo standardized testing to evaluate physical function, cognitive function, and psychiatric function. Added April 2016: They will also undergo a standardized evaluation of speech, swallow, and pain.

ELIGIBILITY:
Inclusion Criteria: Wake Forest MICU Admission

* sepsis OR
* respiratory failure requiring >24 hrs of invasive mechanical ventilation
* previously functional

Exclusion Criteria:

- Active Malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Wake Forest MICU Survivors
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Physical Function | 6 months
  as measured by the Short Performance Physical Battery

SECONDARY OUTCOMES:
Physical Function | 6 months
  Handgrip strength
Cognitive Function | 6 months
  Montreal Cognitive Assessment
Anxiety/ Depression Screening | 6 months
  Hospital Anxiety and Depression Scale
Post Traumatic Stress Disorder Screening | 6 months
  Impact of Events Scale- Revised
Functional Status | 6 months
  Activities of Daily Living and Instrumental Activities of Daily Living
Resilience | 6 months
  Connor-Davidson Resilience Scale- 10
Quality of Life | 6 months
  Short-Form 36
Hospital Readmissions | 6 months
Mortality | 6 months

OTHER OUTCOMES:
Swallow Function | 6 months
  EAT 10 Questionnaire
Speech | 6 months
  Voice Analysis
Pain | 6 months
  Brief Pain Inventory, modified version of the modified musculoskeletal questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: D. Clark Files, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided